CLINICAL TRIAL: NCT00257452
Title: A Double-blind, Randomised, Placebo Controlled, Three-way Cross-over Study With an Open Label Positive Control (Moxifloxacin) to Assess the Influence of Inhaled Tiotropium Once Daily Over Twelve Days on the QTC Interval of the ECG in Healthy Male and Female Volunteers
Brief Title: A Double-blind, Randomised Study to Assess the Influence of Tiotropium (Spiriva®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.302
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tiotropium Bromide; Moxifloxacin

INTERVENTIONS:
Drug: tiotropium 18 mcg or 54 mcg qd
Drug: placebo matching tiotropium qd
Drug: moxifloxacin 200 mg

SUMMARY:
To demonstrate that tiotropium (Spiriva®) does not prolong the QT interval of the ECG more than placebo

DETAILED DESCRIPTION:
The objective of this study is to demonstrate that tiotropium does not prolong the QT interval more than placebo. This will be achieved by testing non-inferiority hypothesis.

Study Hypothesis:

There is one primary variable to be tested for non-inferiority: tiotropium high dose compared to placebo:

H0: µ(TIO,12) - µ(PBO,12) >= 10 ms vs. H1: µ(TIO,12) - µ(PBO,12) < 10 ms where µ(TIO,12), µ(PBO,12) represent the mean change from baseline QTcF between 5 minutes and 2 hours after 12 days of treatment (taking the mean of the time-matched differences between baseline and post-baseline values in each treatment period) with tiotropium 54 µg, or placebo, respectively.

If the data suggest that the Fridericia correction is poor for the study population, an alternative correction will be explored (QTcN). The other correction formula would be used as a replacement for the Fridericia correction and would be defined before unblinding of the data.

Comparison(s):

Placebo, moxifloxacin as active control

ELIGIBILITY:
All participants in the study should be healthy males or females, ranging from 21 to 50 years of age and their body mass index (BMI) be within 18.5 to 29.9 kg/m2 (BMI calculation: weight in kilograms divided by the square of height in meters). In accordance with GCP and the local legislation all volunteers will have given their written informed consent prior to admission to the study.

Exclusion criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug ( two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to tiotropium, moxifloxacin and/or related drugs of these classes
* Heart rate at screening of > 80 bpm or < 45 bpm
* Any screening ECG value outside of the reference range of clinical relevance including, but not limited to PR interval > 220 ms, QRS interval > 115 ms, QTcB or QTcF > 450 ms, or QT (uncorrected) > 470 ms

For Female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilisation, IUP, oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period Lactation period.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Start 2004-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07

PRIMARY OUTCOMES:
Mean change from baseline of the corresponding QTcF values of all ECGs taken from 5 minutes to 2 hours after dosing | Day 12

SECONDARY OUTCOMES:
Mean change from baseline of the corresponding QTcF values of all ECGs taken from 5 minutes to 2 hours after dosing | Day 1
Mean change from baseline of the corresponding QTcF values of all ECGs taken from 5 minutes to 24 hours after dosing | Day 1 and 12
Difference (tiotropium minus placebo) between the maximal time-matched change from baseline of the QTcF values of all ECGs taken from 0:05 - 23:50 after dosing | Day 1 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (1):
- Humanpharmakologisches Zentrum, Ingelheim/Rhein, Germany